CLINICAL TRIAL: NCT03667482
Title: A Phase 1 Study of Concurrent Cabozantinib and Cetuximab in Recurrent or Metastatic Head and Neck Squamous Cell Cancer
Brief Title: Cabozantinib in Combination With Cetuximab in Patients With Recurrent or Metastatic Head and Neck Squamous Cell Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-303
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Head and Neck Squamous Cell Cancer; Recurrent Head and Neck Squamous Cell Cancer; Metastatic Head and Neck Squamous Cell Cancer
Keywords: Cabozantinib; Cetuximab; 18-303
MeSH Terms: interventions — cabozantinib; Cetuximab

STUDY DESIGN:
Intervention Model Description: A standard 3+3 design will be used to find the maximum tolerated dose (MTD) from 3 testing dose levels: 20, 40, and 60.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cabozantinib in Combination With Cetuximab (Experimental): Cetuximab will be administered at 500 mg/m^2 intravenously every other week. Cabozantinib will be initiated at 40 mg PO daily, with subsequent 20 mg or 40 mg doses as tolerated per the study design.
  Interventions: Drug: Cabozantinib; Drug: Cetuximab

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib will be initiated at 40 mg PO daily, with subsequent 20 mg or 40 mg doses as tolerated per the study design.
Drug: Cetuximab — Cetuximab will be administered at 500 mg/m^2 intravenously every other week on Days 1 and 15 of each cycle, with a window of up to 3 days before the scheduled date. In an effort to prevent a hypersensitivity reaction, it is recommended that all patients pre-medications, hydration, and anti-emetics will be given according to institutional guidelines and/or per treating physician discretion.

SUMMARY:
The purpose of this study is to test the safety of cabozantinib, at different doses, in combination with cetuximab to find out what effects, if any, this combined treatment has on people with HNSCC.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet each of the following criteria will be considered "eligible":

* Histologically or cytologically confirmed diagnosis of squamous cell carcinoma of the head and neck.
* Disease must be considered incurable. Incurable is defined as metastatic disease or a local or regional recurrence in a previously irradiated site that is unresectable (or patient declines resection).
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >10 mm with CT scan, as >20 mm by chest x-ray, or >10 mm with calipers by clinical exam.
* Patients may have received pembrolizumab, platins, cetuximab or other chemotherapies in the metastatic setting, but do not need to have received cetuximab.
* Measurable disease per RECIST v1.1 as determined by the investigator;
* The subject has had an assessment of all known disease sites e.g., by computerized tomography (CT) scan, magnetic resonance imaging (MRI), bone scan as appropriate, within 28 days before the first dose of cabozantinib.
* A CT of the neck and a CT of the chest will be required at baseline for all patients.
* The subject is ≥ 18 years old on the day of consent.
* The subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Recovery to baseline or ≤ Grade 1 CTCAE v.5.0 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy.
* The subject has organ and marrow function and laboratory values as follows within 14 days before the first dose of cabozantinib.

  1. The ANC ≥ 1500/mm3 without colony stimulating factor support.
  2. White blood cell count ≥ 2500/mm3 (≥ 2.5 GI/L).
  3. Platelets ≥ 100,000/mm3;
  4. Hemoglobin ≥ 9 g/dL;
  5. Bilirubin ≤ 1.5 x the ULN. For subjects with known Gilbert's disease, bilirubin ≤ 3.0 mg/dL;
  6. Albumin ≥ 2.8 g/dl;
  7. Creatinine ≤ 2.0 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min. For creatinine clearance estimation, the Cockcroft and Gault equation should be used:

  i. Male: CrCl (mL/min) = (140 - age) × wt (kg) / (creatinine × 72); h. Female: Multiply above result by 0.85; Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) ≤ 3 x upper limit of normal (ULN). ALP ≤ 5 x ULN with documented bone metastases.

  i. Lipase < 2.0 x the upper limit of normal and no radiologic or clinical evidence of pancreatitis.

  j. UPCR ≤ 1. k. Phosphorus, calcium, magnesium and potassium ≥ LLN.
* The subject is capable of understanding and complying with the protocol requirements and has signed the informed consent document;
* Sexually active subjects (men and women) must agree to use medically accepted barrier methods of contraception (e.g., male or female condom) during the course of the study and for 4 months after the last dose of study drug(s), even if oral contraceptives are also used. All subjects of reproductive potential must agree to use both a barrier method and a second method of birth control during the course of the study and for 4 months after the last dose of study drug(s).
* Female subjects of childbearing potential must not be pregnant at screening. Females of childbearing potential are defined as premenopausal females capable of becoming pregnant (i.e., females who have had any evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy). However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, low body weight, ovarian suppression or other reasons.
* No Grade 3-4 hypersensitivity reaction to cetuximab.

Exclusion Criteria:

Patients who meet any of the following criteria will be considered "ineligible":

* Any patient who has received >70 Gy of XRT to the neck in the same radiation field. No head and neck radiation within 2 months prior to initiation. Treatment areas should be healed with no sequelae from RT that would predispose to fistula formation.
* A history of other malignancy ≤ 5 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only, carcinoma in situ of the cervix, synchronous H&N primaries or low grade tumors deemed cured and not treated with systemic therapy. Other cancers that will not affect the study outcome may be included with the consent of the PI (Dr. Michel) as long as it would not affect the study outcome (e.g., low grade prostate cancer on surveillance alone).
* Receipt of any type of cytotoxic, biologic or other systemic anticancer therapy (including investigational) within 4 weeks before first dose of study treatment with the exception of cetuximab and small molecule kinase inhibitors (kinase inhibitors must be stopped within 2 weeks of first dose of study treatment.
* Prior treatment with cabozantinib.
* Radiation therapy for bone metastasis within 2 weeks, any other external radiation therapy within 4 weeks before the first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before the first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.;
* Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 14 days before the first dose of study treatment. Note: Subjects with prostate cancer currently receiving LHRH or GnRH agonists may be maintained on these agents.
* The subject has received any other type of investigational agent within 28 days before the first dose of study treatment.
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before the first dose of study treatment. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of the start of study treatment.
* The subject has prothrombin time (PT)/INR or partial thromboplastin time (PTT) test ≥ 1.3 x the laboratory ULN within 7 days before the first dose of study treatment.
* Concomitant anticoagulation with oral anticoagulants (e.g., warfarin, direct thrombin and Factor Xa inhibitors) or platelet inhibitors (e.g., clopidogrel).

Allowed anticoagulants are the following:

1. Low-dose aspirin for cardioprotection (per local applicable guidelines) is permitted.
2. Low-dose low molecular weight heparins (LMWH) are permitted.
3. Anticoagulation with therapeutic doses of LMWH is allowed in subjects without known brain metastases who are on a stable dose of LMWH for at least 6 weeks before first dose of study treatment, and who have had no clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.

   * The subject has experienced any of the following:

a. clinically-significant GI bleeding within 6 months before the first dose of study treatment; b. hemoptysis of ≥ 0.5 teaspoon (2.5ml) of red blood within 3 months before the first dose of study treatment;

* Any other signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment. Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 12 weeks before first dose.
* Cavitary lesions <=4cm are allowed unless they are abutting major vessels. Patients with pleural-based lesions will be closely monitored for signs of pneumothorax by chest XR or CT if acute shortness of breath is reported or other signs/symptoms of hypoxia are apparent.
* The subject has tumor invading or encasing any major blood vessels.
* The subject has evidence of tumor invading the GI tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of cabozantinib.
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before the first dose of study treatment. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of the start of study treatment.
* The subject has prothrombin time (PT)/INR or partial thromboplastin time (PTT) test ≥ 1.3 x the laboratory ULN within 7 days before the first dose of study treatment.
* Concomitant anticoagulation with oral anticoagulants (e.g., warfarin, direct thrombin and Factor Xa inhibitors) or platelet inhibitors (e.g., clopidogrel). Allowed anticoagulants are the following:

  1. Low-dose aspirin for cardioprotection (per local applicable guidelines) is permitted.
  2. Low-dose low molecular weight heparins (LMWH) are permitted.
  3. Anticoagulation with therapeutic doses of LMWH is allowed in subjects without known brain metastases who are on a stable dose of LMWH for at least 6 weeks before first dose of study treatment, and who have had no clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.
* The subject has experienced any of the following:

  1. clinically-significant GI bleeding within 6 months before the first dose of study treatment;
  2. hemoptysis of ≥ 0.5 teaspoon (2.5ml) of red blood within 3 months before the first dose of study treatment;
* any other signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment. Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 12 weeks before first dose.
* The subject has radiographic evidence of cavitating pulmonary lesion(s).
* The subject has tumor invading or encasing any major blood vessels.
* The subject has evidence of tumor invading the GI tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of cabozantinib.
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  a. Cardiovascular disorders including: i. Congestive heart failure (CHF): New York Heart Association (NYHA) Class III (moderate) or Class IV (severe) at the time of screening; ii. Concurrent uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mm Hg systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment within 7 days of the first dose of study treatment; iii. Any history of congenital long QT syndrome; iv. Any of the following within 6 months before the first dose of study
  * treatment: unstable angina pectoris;
  * clinically-significant cardiac arrhythmias;
  * stroke (including transient ischemic attack (TIA), or other ischemic event);
  * myocardial infarction;
  * thromboembolic event requiring therapeutic anticoagulation (Note: subjects with a venous filter (e.g., vena cava filter) are not eligible for this study).
* GI disorders particularly those associated with a high risk of perforation or fistula formation including: i. Tumors invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (e.g., Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction. Abdominal fistula, GI perforation, bowel obstruction, intra-abdominal abscess within 6 months before randomization

  * Note: Complete healing of an intra-abdominal abscess must be confirmed prior to randomization ii.

ii. No pre-existing fistula of the head and neck. No pre-existing osteonecrosis of the jaw.

* Other clinically significant disorders that would preclude safe study participation;
* Major surgery (e.g., GI surgery, removal or biopsy of brain metastasis) within 8 weeks before first dose of study treatment. Complete wound healing from major surgery must have occurred 1 month before first dose and from minor surgery (e.g., simple excision, tooth extraction) at least 10 days before first dose. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 msec within 1 month before the first dose of study treatment:

  a. If a single ECG shows a QTcF with an absolute value > 500 ms, two additional ECGs must be performed within 30 minutes after the initial ECG, and the average of these three consecutive results for QTcF will be used to determine eligibility.
* Pregnant or lactating females;
* Inability to swallow intact tablets;
* Previously identified allergy or hypersensitivity to components of the study treatment formulations;
* The subject requires chronic concomitant treatment with strong CYP3A4 inducers (e.g., phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital, and St.

John's Wort).

* Other clinically significant disorders that would preclude safe study participation.

  1. Serious non-healing wound/ulcer/bone fracture.
  2. Symptomatic hypothyroidism.
  3. Moderate to severe hepatic impairment (Child-Pugh B or C).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) | 2 years
  from 3 testing dose levels: 20, 40, and 60. Three patients will be enrolled at the dose level 0 of 40 mg. The dose escalation scheme is as follows:
  1. If none of the initial three patients at a given dose level experience DLT within 4 weeks, the next dose level will be studied.
  2. If one of the initial three patients at a given dose level experiences DLT, three additional patients will be treated at the same dose level. Escalation will continue only if there is no additional DLT observed.If two or more patients experience DLT at a given dose, the previous dose level will be studied. Should two or more patients experience the DLT at the lowest dose level (20 mg), the study will be halted, and alternative dosing will be considered.
  4. The highest dose level with no more than one DLT among six patients will be declared as the MTD. If only three patients were treated at a dose under consideration as the MTD, an additional three patients will be treated at that level.

CONTACTS AND LOCATIONS:
Overall Officials: Loren Michel, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - Baptist Alliance MCI, Miami, Florida
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Lehigh Valley Health Network, Allentown, Pennsylvania

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm